CLINICAL TRIAL: NCT05799053
Title: Peppermint Oil for the Treatment of Irritable Bowel Syndrome or Functional Abdominal Pain in Children: the MINT Study
Acronym: MINT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: St. Antonius Hospital (Other)
Responsible Party: Principal Investigator, Koen Vermeijden, MD, St. Antonius Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NL78304.100.21
Record Dates: First submitted 2023-02-07; First posted 2023-04-05 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2024-04

CONDITIONS: Irritable Bowel Syndrome; Functional Abdominal Pain Syndrome; Child; Adolescent; Therapeutics; Adverse Drug Event
Keywords: Peppermint oil; Irritable Bowel Syndrome; Functional Abdominal Pain - Not Otherwise Specified; Paediatrics
MeSH Terms: conditions — Irritable Bowel Syndrome; Drug-Related Side Effects and Adverse Reactions | interventions — peppermint oil

STUDY DESIGN:
Intervention Model Description: Patients are randomized in three groups: 1) peppermint oil capsules, 2) placebo), peppermint sweets
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Peppermint oil capsules and placebo are double blinded, peppermint sweets are open-label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Peppermint oil capsules (Tempocol®) (Experimental): Enteric-coated capsule containing 182mg of Peppermint Oil that release the oil in the small intestine, to be taken orally.
  Age: 8-11 years old: 2 times daily for 8 weeks, if needed upped to 3 times daily after 4 weeks Age: 12-18: 3 times daily for 8 weeks, if needed upped to 3 times two capsules daily after 4 weeks
  Interventions: Drug: Small intestinal release peppermint oil
- Placebo (Placebo Comparator): Capsule containing microcrystalline cellulose, to be taken orally. Age: 8-11 years old: 2 times daily for 8 weeks, if needed upped to 3 times daily after 4 weeks Age: 12-18: 3 times daily for 8 weeks, if needed upped to 3 times two capsules daily after 4 weeks
  Interventions: Drug: Placebo
- Peppermint sweets (Wilhelmina®) (Experimental): Wilhelmina® peppermints contain 9.2 mg of Menthae Piperitae Aetheroleum (peppermint oil), and 18.4 Kcal per mint and are to be taken orally.
  Age: 8-11 years old: 2 times daily for 8 weeks, if needed upped to 3 times daily after 4 weeks Age: 12-18: 3 times daily for 8 weeks, if needed upped to 3 times two capsules daily after 4 weeks
  Interventions: Drug: Peppermint sweets

INTERVENTIONS:
Drug: Small intestinal release peppermint oil — Tempocol®, a gastric acid resistant (enteric-coated) capsule containing 182mg of Menthae Piperitae Aetheroleum (peppermint oil), is currently registered as an over the counter prescription drug on the Dutch market for treatment of abdominal pain, discomfort or flatulence.
  Other Names: Peppermint oil; Menthae piperitae aetheroleum; Tempocol®; A03AX15
  Arms: Peppermint oil capsules (Tempocol®)
Drug: Peppermint sweets — Wilhelmina® peppermints contain 9.2 mg of Menthae Piperitae Aetheroleum (peppermint oil), and 18.4 Kcal per mint and are to be taken orally.
  Other Names: Wilhelmina®
  Arms: Peppermint sweets (Wilhelmina®)
Drug: Placebo — Capsule containing microcrystalline cellulose
  Arms: Placebo

SUMMARY:
Peppermint oil has shown to be effective in the treatment of Irritable Bowel Syndrome (IBS) symptoms in adults. Few studies of low quality are performed in an paediatric setting. Therefore, the investigators will conduct a multicenter randomized, placebo controlled trial to investigate the effects of an eight-week peppermint oil treatment in paediatric IBS or Functional Abdominal Pain - Not otherwise specified (FAP-NOS) patients.

DETAILED DESCRIPTION:
The objective of the MINT study is to investigate the effectiveness of peppermint oil capsules compared to placebo capsules in reducing abdominal pain intensity in children with IBS or FAP-NOS. In addition, we evaluate the effect of peppermint oil capsules compared to placebo capsules on other disease-related outcome measures such as anxiety & depression, quality of life, absenteeism from school, and healthcare costs. The second aim is to explore the effectiveness of regular mints in reducing abdominal pain intensity compared to peppermint oil capsules and placebo capsules and the effect of mints on secondary outcome parameters.

ELIGIBILITY:
Inclusion Criteria:

* Children aged between 8 years and 18 years
* Diagnosis of IBS or FAP-NOS according to the Rome IV criteria. According to these criteria, organic disorders will be ruled out after routine laboratory testing initiated by their general practitioner or treating physician as part of standard of care. In patients without alarm symptoms only celiac screening (anti-transglutaminase antibodies and IgA), and faecal calprotectin are necessary.37 In patients with diarrhea faecal testing for Giardia Lambliae will be added. If alarm symptoms are present, further diagnostic testing (like a full blood count, CRP, liver tests or an ultrasound) to rule out an organic disorder, is left to the discretion of the treating physician.
* An average daily pain rate of ≥ 3 of 10 on the Wong Baker Faces Pain Scale (This is a validated pain scale to measure pain intensity).

Informed Consent by both parents and by children aged ≥ 12 years. No informed consent from parents is necessary for children >16 years.

Exclusion Criteria:

* Current treatment by another health care professional for abdominal symptoms
* Previous use of peppermint oil for these abdominal complaints
* Known hypersensitivity to mints or peppermint oil
* Gastrointestinal blood loss
* Recurrent or unexplained fevers
* Decreased growth velocity
* History of previous abdominal surgeries in the past 3 months
* Significant chronic health condition requiring specialty care (e.g., lithiasis, ureteropelvic junction obstruction, sickle cell, cerebral palsy, hepatic, hematopoietic, renal, endocrine, or metabolic diseases) that could potentially impact the child's ability to participate or confound the results of the study
* Known concomitant organic gastrointestinal disease
* Current use of drugs which influence gastrointestinal motility, such as erythromycin, azithromycin, butyl scopolamine, domperidone, mebeverine and Iberogast. If laxatives are being used (in patients with IBS-C) they can continue using them during the study.
* Current use of proton-pump inhibitors
* Insufficient knowledge of the Dutch language
* Pregnancy or current lactation. Women with childbearing potential must have a negative urine pregnancy test within 7 days prior to first dose of study treatment

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 228 (Actual)
Dates: Start 2022-05-12 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Abdominal pain intensity response rate after 8 weeks of treatment | 8 weeks
  The proportion of patients with ≥ 30% reduction of their abdominal pain intensity after 8 weeks of therapy compared to baseline. This will be assessed by a smartphone diary app, on which patients record daily at the end of the day the intensity of their abdominal pain during a period of 7 consecutive days using a 10 point Likert scale/Wong-Baker faces scale. A score of 0 correlates with no pain and a score of 10 correlates with the worst imaginable pain. The intensity scores of 7 days will be summed up.

SECONDARY OUTCOMES:
Change in pain duration | 4 weeks, 8 weeks, 12 weeks
  Abdominal pain duration will be scored in minutes of abdominal pain per day during 7 consecutive days after 8 weeks of therapy compared to baseline
Change in pain frequency | 4 weeks, 8 weeks, 12 weeks
  Abdominal pain frequency will be scored as the average amount of days with pain during 7 consecutive days after 8 weeks of therapy compared to baseline
Change in abdominal pain intensity | 4 weeks, 8 weeks, 12 weeks
  Abdominal pain intensity will be scored using a 10-point Wong-Baker faces scale during 7 consecutive days after 8 weeks of therapy compared to baseline
Change in Quality of Life | 8 weeks
  Change in quality of live will be measured with the PedsQL after 8 weeks of therapy compared to baseline
Change in depression and anxiety score | 8 weeks
  Depression and anxiety scores are measured by the Revised Anxiety and Depression Scale-short version (RCADS-25) after 8 weeks of therapy compared to baseline
School absences during the treatment | 4 weeks, 8 weeks, 12 weeks
  Hours of school absence in the previous week are measured.
Use of pain rescue medication during the treatment | 4 weeks, 8 weeks, 12 weeks
  Use of pain rescue medication like paracetamol or NSAIDs
Expectancy of treatment | 0 weeks
  expectations of both parents separately of the treatment on a scale of 0 (no improvement) to 10 (very much improved)
Expectancy of treatment | 0 weeks
  the child's expectations of the treatment on a scale of 0 (no improvement) to 10 (very much improved)
Change in defecation pattern | 4 weeks, 8 weeks, 12 weeks
  Change in defecation pattern is recorded as the daily stool frequency and consistency according to the Bristol Stool Scale
Adequate relief | 4 weeks, 8 weeks, 12 weeks
  patients will be asked whether they have adequate relief of IBS/FAP-NOS symptoms using a single question ("Did you have adequate relief of IBS/FAP-NOS symptoms (abdominal discomfort/pain, bowel habits, and other symptoms like nausea and bloating) over the past week?") scored on a dichotomous scale (Yes/No)
Health status | 8 weeks
  the EQ-5D-Y is a standardised questionnaire on health-related quality of life and will be used in the cost-effectiveness and cost-utility analysis
Costs | 8 weeks, 12 weeks
  iMCQ and the iPCQ will be used to measure the direct and indirect costs due to health care utilization and work absenteeism by parents
Safety of peppermint oil | 4 weeks, 8 weeks, 12 weeks
  incidence of adverse events will be reported by the participants
Ease of use of peppermint oil capsules, placebo capsules or peppermint sweets | 8 weeks
  Ease of use of capsules or sweets will be scored after 8 weeks using a 5-point Likert scale with the following statement: the pills were easy to use and swallow: strongly disagree/disagree/neither agree nor disagree/agree/strongly agree.
Taste of peppermint oil capsules, placebo capsules or peppermint sweets | 8 weeks
  taste of capsules or sweets will be scored after 8 weeks using a Likert scale: I like the taste of the pills: strongly disagree/disagree/neither agree nor disagree/agree/strongly agree.
Placebo genes | 0 weeks
  Several other single nucleotide polymorphisms (SNPs) were found to influence response to placebo treatment. Therefore, we will investigate whether SNPs in a candidate set of genes (previously associated with either the placebo response in adults) are related to either placebo response or treatment response in children with IBS or FAP-NOS.

CONTACTS AND LOCATIONS:
Overall Officials: Arine Vlieger, MD, PhD, Principal Investigator — St. Antonius Hospital
Locations (3):
- Netherlands (3):
  - De KinderKliniek, Almere Stad, Flevoland
  - Amphia Hospital, Breda, North Brabant
  - Amsterdam UMC, Amsterdam, North Holland